CLINICAL TRIAL: NCT04877132
Title: Compassionate Use Program for Olipudase Alfa Enzyme Replacement Therapy for Patients With Chronic Acid Sphingomyelinase Deficiency (ASMD)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: RHASHC09706
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Sphingomyelin Lipidosis
MeSH Terms: conditions — Niemann-Pick Disease, Type A | interventions — olipudase alfa

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: olipudase alfa (GZ402665) — Patients will receive intravenous (IV) infusion of olipudase alfa

SUMMARY:
The objective of this program is to provide access to enzyme replacement therapy (ERT) with olipudase alfa for certain patients with ASMD, a severe, life threatening disease, that could not participate in the olipudase clinical trials. The program will provide access to olipudase alfa prior to registration and the availability of commercial product (including reimbursement where applicable) in the country of the patient.

ELIGIBILITY:
Inclusion Criteria:

All patients (adult and pediatric)

* Unsolicited request for the patient from a site with at least 3 years of experience in administration and safety management of ERT.
* Written informed consent signed by the patient or the patient's parent(s)/guardian(s), where applicable.
* Documented deficiency of acid sphingomyelinase in peripheral leukocytes, lymphocytes, or cultured fibroblasts.

Adult patients

* Age ≥ 18 years.
* Clinically documented advanced disease evidenced by defined thresholds for lung, spleen, liver, and hematologic parameters.

Pediatric patients

- Age >3 years and <18 years or clinical diagnosis consistent with ASMD Type A/B or Type B.

Exclusion Criteria:

All patients (adult and pediatric)

* Active serious intercurrent illness which will preclude enrollment, significant liver disease with etiology other than ASMD, Malignancy with poor prognosis, serious medical or psychiatric condition that may preclude participation, or circumstances that may interfere with compliance in this compassionate use program, requirement for recurrent dose adjustment of anticoagulation treatment over the last 6 months.
* Pregnancy or breastfeeding.
* For female patients of childbearing potential, a positive serum pregnancy (β human chorionic gonadotropin [HCG]) test result.
* For female patients of childbearing potential and sexually active male patients, unwillingness to abstain from heterosexual intercourse in accordance with their preferred and usual lifestyle, or to use 2 acceptable, effective contraceptive methods, while participating in this program and for 15 days after the last infusion of olipudase alfa.
* For pediatric patients, clinical diagnosis, or suspicion of infantile onset ASMD. Genotype compatible with ASMD type A.

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi